CLINICAL TRIAL: NCT03856619
Title: A Single Arm Phase IV Clinical Trial to Describe the Safety and Efficacy of Teriflunomide in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: To Evaluate the Safety and Efficacy of Teriflunomide in Patients With Relapsing Forms of Multiple Sclerosis
Acronym: SAFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TERIFL08918; U1111-1205-3009 (Other: UTN)
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — teriflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aubagio®/Teriflunomide (Experimental): Single dose of Aubagio® to be taken orally, once daily in the morning
  Interventions: Drug: TERIFLUNOMIDE HMR1726

INTERVENTIONS:
Drug: TERIFLUNOMIDE HMR1726 — Pharmaceutical form: Tablet
  Route of administration: Oral

SUMMARY:
Primary Objective:

To describe the safety of teriflunomide in patients with relapsing forms of multiple sclerosis.

Secondary Objective:

To describe the efficacy of teriflunomide in patients with relapsing forms of multiple sclerosis.

DETAILED DESCRIPTION:
The study duration is one year; post treatment safety follow up visit will be conducted 4 weeks after the patient takes the last dose of teriflunomide

ELIGIBILITY:
Inclusion criteria:

* Age of patients ≥ 18 years
* Patients with relapsing form of multiple sclerosis at time of screening visit.
* Signed written informed consent.

Exclusion criteria:

* Patients with hypersensitivity to teriflunomide, leflunomide, or to any excipients in the tablets.
* Liver function impairment or persisting elevations of serum glutamic pyruvic transaminase (SGPT/ALT), serum glutamic oxaloacetic transaminase (SGOT/AST), greater than two times the upper limit of normal (ULN) during screening visit.
* Known history of pre-existing acute or chronic liver disease.
* Patients with significantly (as per Investigator's discretion) impaired bone marrow function or significant anemia, leukopenia, or thrombocytopenia.
* Known history of severe immunodeficiency, acute or severe active infections.
* Female patients with a positive pregnancy test at screening or women of child-bearing potential who do not agree to use effective methods of contraception throughout the course of the study.
* Male patients unwilling to use reliable contraception during the course of the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | 1 year
  Incidence of adverse events

SECONDARY OUTCOMES:
Annualized relapse rate | 1 year
  Number of relapses per patient-year
First relapse | 1 year
  Time to first relapse
Relapse free | 1 year
  Proportion of patients who are relapse free
Neurological impairment/disability | Baseline to 3 months, 6 months, 9 months and 1 year
  Expanded Disability Status Scale (EDSS) will be used to compare disability from baseline. The EDSS ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Disability progression | 1 year
  Proportion of patients free of disability progression
Drug compliance | 1 year
  Percentage of patients who are treatment compliant assessed using patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- India (14):
  - Investigational Site Number :024, Ahmedabad
  - Investigational Site Number :017, Bengaluru
  - Investigational Site Number :001, Chandigarh
  - Investigational Site Number :023, Coimbatore
  - Investigational Site Number :007, Gūrgaon
  - Investigational Site Number :026, Gūrgaon
  - Investigational Site Number :005, Kochi
  - Investigational Site Number :006, Kolkata
  - Investigational Site Number :011, Lucknow
  - Investigational Site Number :020, Ludhiana
  - Investigational Site Number :018, Nashik
  - Investigational Site Number :025, New Delhi
  - Investigational Site Number :014, Pune
  - Investigational Site Number :022, Thiruvananthapuram

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.clinicalstudydatarequest.com/